CLINICAL TRIAL: NCT03767816
Title: The Visceral Analgesic Effect of Erector Spinae Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hyuk Lee, clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-1320
Record Dates: First submitted 2018-11-15; First posted 2018-12-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Visceral Pain, Postoperative
Keywords: laparoscopic cholecystectomy; erector spinae plane block; visceral pain
MeSH Terms: conditions — Visceral Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R : Rectus sheath block group (Experimental): ultrasound guided Rectus sheath block with 0.2% ropivacaine (Fresenius Kabi) 30ml before surgical incision
  Interventions: Drug: Ultrasound guided Rectus sheath block
- Group RE: Rectus sheath block and erector spinae plane block (Active Comparator): ultrasound guided Rectus sheath block with 0.2% ropivacaine (Fresenius Kabi) 30ml before surgical incision and ultrasound guided erector spinae plane block with 0.2% ropivacaine (Fresenius Kabi) 40ml
  Interventions: Drug: Ultrasound guided Rectus sheath block; Drug: Ultrasound erector spinae plane block

INTERVENTIONS:
Drug: Ultrasound guided Rectus sheath block — Ultrasound guided rectus sheath block with 0.2% ropivacaine (Fresenius Kabi) 30ml around umbilicus
Drug: Ultrasound erector spinae plane block — Ultrasound guided erector spinae plane block with 0.2% ropivacaine (Fresenius Kabi) 40ml at T7 level
  Arms: Group RE: Rectus sheath block and erector spinae plane block

SUMMARY:
The purpose of this study was to investigate the effectiveness of erector spinae plane block on postoperative visceral pain in laparoscopic cholecystectomy (LLC). Given that rectus sheath block may provide sufficient somatic pain block, investigators aimed to investigate whether erector spinae block is effective in visceral pain block.

After induction of general anesthesia, group of patient is decided randomly. In Group R, rectus sheath block is performed with 0.2% Ropivacaine 30ml before the operation. In Group RE, rectus sheath block and erector spinae plane block are performed with 0.2% ropivacaine 70ml before the operation.

NRS score measurement and comparison of the rescue analgesic dose used at 0, 0.5, 1, 2,6, 12, 18, and 24 hours after arrival at the recovery room were collected

ELIGIBILITY:
Inclusion Criteria:

1. adults between the ages of 20 and 80
2. scheduled laparoscopic cholecystectomy patient
3. American society of anesthesiologists score 1 or 2
4. Patients who have voluntarily agreed in writing to participate in the trial

Exclusion Criteria:

1. Patient with side effects on local anesthetics or steroids
2. Patient who are taboo of peripheral nerve block such as blood clotting disorder, infection, etc.
3. Patients with uncontrolled medical or psychiatric problem
4. Patient does not agree to participate in the study
5. Patients with deformity at vertebra or chest wall.
6. Patients who are pregnant or lactating
7. Patients receiving a single laparoscopic cholecystectomy (including using a robot)
8. Patients with severe intraperitoneal adhesion (higher than Nair s grade 3), or with external drain.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Difference of analgesic consumption between both group | at 0, 0.5, 1, 2, 6, 12, 18, 24 hours after operation
  The difference in analgesics usage between the two groups after the operation is checked at fixed intervals (at 0, 0.5,
  1, 2, 6, 12, 18, 24 hours after operation) to compare.

SECONDARY OUTCOMES:
compare the Numeric rating scale (NRS) | at 0, 0.5, 1, 2, 6, 9, 18, 24 hours after operation
  10 years old or older. 0: No pain, 1-3: mild pain, 4-6: Moderate pain, 7-10: severe pain, 10: worst pain imaginable.
  After surgery, the NRS differences between the two groups were compared at a constant interval (0, 0.5, 1, 2, 6, 12, 18, 24 hours postoperatively).

CONTACTS AND LOCATIONS:
Overall Officials: JongHyuk Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea